CLINICAL TRIAL: NCT01307839
Title: A Randomized, Controlled Trial of the Lidocaine Patch for Relief of Pain During Epidural Needle Insertion in Laboring Patients
Brief Title: Lidocaine Patch for Relief of Pain During Epidural Placement in Laboring Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to non-availability of the lidocaine placebo patches.
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Richard Applegate, MD, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5110014
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Pregnant; Labor
Keywords: labor; epidural

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5% lidocaine patch (Active Comparator): If the patient chooses to participate, the resident will place the patch over the lower lumbar area of the back.
  Interventions: Drug: 5% lidocaine patch
- placebo patch (Placebo Comparator): If the patient chooses to participate, the resident will place the patch over the lower lumbar area of the back.
  Interventions: Drug: placebo patch

INTERVENTIONS:
Drug: 5% lidocaine patch — Research intervention: After consent has been given, either an active 5% lidocaine patch or an inactive placebo patch will be placed on the lumbar spine of the patient. Both patches appear identical to the physician. The team will then wait for the patient to request an epidural due to labor pain, a minimum of 30 minutes from patch placement and a maximum of 12 hours.
  Arms: 5% lidocaine patch
Drug: placebo patch — Research intervention: After consent has been given, either an active 5% lidocaine patch or an inactive placebo patch will be placed on the lumbar spine of the patient. Both patches appear identical to the physician. The team will then wait for the patient to request an epidural due to labor pain, a minimum of 30 minutes from patch placement and a maximum of 12 hours
  Arms: placebo patch

SUMMARY:
Infiltration of the skin with lidocaine is standard practice prior to lumbar epidural placement in laboring parturients1. Skin infiltration, although brief, can be very stressful and painful for patients.2 This initial discomfort may cause patient anxiety, thus increasing the pain and decreasing the satisfaction with the procedure. To reduce this discomfort, various topical alternatives have been investigated with varying degrees of success.1-4 Now that a topical mixture of lidocaine that is safe and effective is available, the investigators would like to determine if it can reduce the pain of skin infiltration in particular and epidural placement as a whole.

ELIGIBILITY:
Inclusion Criteria:

1. Laboring patients between the ages of 18 and 45 with a BMI of less than 45

Exclusion Criteria:

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
To determine if the 5% lidocaine patch can decrease the pain from epidural placement. | a minimum of 30 minutes from patch placement and a maximum of 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Applegate, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States